CLINICAL TRIAL: NCT03916653
Title: Clinical and Radiographic Comparative Evaluation of Osseous Resection by Piezoelectric Device Versus Conventional Rotary Instruments in Crown Lengthening Procedure: A Randomized Controlled Clinical Trial
Brief Title: Comparative Evaluation of Osseous Resection by Piezoelectric Device Versus Conventional Rotary Instruments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: prinita perio
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-04

CONDITIONS: Healing Surgical Wounds

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Osseous resection using piezoelectric device
  Interventions: Procedure: osseous resection using piezoelectric device in surgical crown lengthening
- Control group (Active Comparator): Osseous resection using conventional rotary instruments
  Interventions: Procedure: Osseous resection using conventional rotary instruments in surgical crown lengthening

INTERVENTIONS:
Procedure: osseous resection using piezoelectric device in surgical crown lengthening — In this group piezoelectric device will be used for osseous resection in crown lengthening procedure with copious irrigation of sterile saline.
  Arms: Test group
Procedure: Osseous resection using conventional rotary instruments in surgical crown lengthening — For osseous resection in crown lengthening procedure, conventional rotary instruments will be used with copious irrigation of sterile saline.
  Arms: Control group

SUMMARY:
The aim of this study is to comparatively evaluate changes in periodontal healing, surgical time required and postoperative morbidity observed in patients undergoing osseous resection in crown lengthening procedure with conventional rotary instruments versus piezoelectric device.

DETAILED DESCRIPTION:
Surgical Crown lengthening (SCL) procedure facilitates restorative and prosthetic rehabilitation to provide adequate clinical crown structure to teeth which are otherwise compromised due to subgingival pathologies. One of the main advantages of the surgery is gain in supragingival crown length which is desirable for restoring severely lost tooth structure. This procedure provides increase in retention and resistance forms of the tooth necessary for restorative treatment. Indications of this procedure are subgingival caries, crown & root fracture, short clinical abutments, cervical root resorption and altered passive eruption.

Gargiulo et al. has given the concept of biologic width the distance between the base of the gingival sulcus and height of alveolar crest) based on classic histologic study in humans. He measured the average dimensions of epithelial junction and connective tissue attachment, the summed value of these dimensions gave biological width (2.04mm=0.97mm+1.07mm). Later on, Vacek et al.2 examined naturally occurring dimensions in human cadaver histomorphometrically and measured mean dimensions for epithelial attachment (1.14 +/- 0.49 mm) and for connective tissue attachment(0.77 +/- 0.32 mm). The average dimensions reported was approximately 2mm. The importance of biologic width lies in the fact that the violation of this width leads to gingival inflammation, attachment loss, and alveolar bone resorption. The integrity of biologic width should be maintained while performing crown lengthening for healthy hard and soft tissues, required for prosthetic and restorative rehabilitations.

Nevins M et al. and Ingber JS et al. proposed "3mm rule" for crown lengthening. According to this, 3mm of alveolar bone should be removed during crown lengthening, but this can not be applicable to all cases. Deas DE et al. in a study demonstrated significant tissue rebound following crown lengthening which was found to be related to placement of flap with respect to alveolar crest. More the distance between POST SUTURING Flap position and alveolar crest, less was the tissue rebound observed.

Osseous surgery in crown lengthening can be performed using rotary & manual instruments like carbide diamond burs, surgical chisels and files which leads to generation of heat, post-operative discomfort, swelling and trismus. Vercellotti et al. proposed that Piezosurgery is a new osteotomy procedure that requires microvibrations at ultrasonic frequency facilitated to cut hard tissue, while soft tissue remained unaffected. The sites treated with piezoelectric device had gain in bone level compared to sites treated by carbide bur or diamond bur. Ma LI et al and Esteves JC et al in a study performed on animals, demonstrated that the use of piezoelectric device in bone cutting showed advanced bone healing compared to traditional bone cutting. Sortino et al. proposed that piezosurgery osteotomy showed less post-operative complications (facial swelling, trismus, discomfort) although it required longer time for surgery. Verardi S.et al. evaluated and proposed that piezosurgery showed more favorable response in periodontal compromised patients in terms of less chewing discomfort, less cold sensitivity and low pain perception at various time points compared to conventional surgical treatment.

Till date, no studies have compared the periodontal healing, patient based perception of pain, and discomfort after osseous resection in crown lengthening using piezosurgery with conventional rotary instruments. The aim of this study is to comparatively evaluate, clinically and radiographically,the changes in periodontal healing, surgical time required and postoperative morbidity observed in patients undergoing osseous resection in crown lengthening procedure with conventional rotary instruments versus piezoelectric device.

The present prospective, analytical, randomized controlled clinical trial will be conducted in the Department of Periodontics and Oral Implantology, Post Graduate Institute of Dental Sciences, Rohtak Systemically healthy patients age group 18-60years will participate in this study. Each patient should have at least one tooth for conducting crown lengthening procedure either in maxillary or mandibular arch.

Participants will be enlisted from the regular outpatient department of the Department of Periodontics and Oral Implantology and Department of Oral Medicine and Radiology after screening on the basis of inclusion and exclusion criteria . All participants will be given an outline of the study design and all patient-specific considerations and concerns will be properly addressed. All participants will be required to provide written informed consent. All patients enrolled in the study will be further randomly divided into the following two groups using computer-generated balanced block randomization table with 1:1 allocation

1. Control group - For osseous resection in crown lengthening procedure, conventional rotary instruments will be used with copious irrigation of sterile saline.
2. Test group-In this group piezoelectric device will be used for osseous resection in crown lengthening procedure with copious irrigation of sterile saline.

Control Group Before surgical procedure all clinical measurements will be recorded using customized acrylic stents and radiograph will be taken. Administration of local anesthesia will be done for nerve block. Incisions will be given based on width of keratinized gingiva. Before resective surgery, the position of free gingival margins (FGM) will be recorded from the stent which will be placed on teeth before surgery, using periodontal probe. Intrasulcular incisions/internal bevel incisions will be given and elevation of full thickness mucoperiosteal flap will be done in both buccal and lingual aspect. The osseous resection will be performed based on presence amount of tooth structure to be gained for future restorative rehabilitation. The ostectomy (removal of bone supporting teeth) will be performed under combination of rotary instruments, bone chisels, carbide & diamond burs with copious saline irrigation & maintenance of natural bone anatomy and architecture throughout the procedure. Exposed root surfaces will be planed to prevent re-attachment and rebounding of free gingival margins to its initial position. After planning, the surgical sites will be closed after applying pressure for 3min and providing adaption. Suturing of flap shall be done based on presence of supracrestal gingival tissues(SGT) acquired postoperatively ,maintaining the preoperative dimensions of the SGT. Fixation of flap then placing apically to ensure maximum facial & lingual bone coverage. Measurements of parameter will be recorded by single investigator before and after surgery and post operative instructions will be given to patients once all procedure is completed. Patients will be recalled after 1week for suture removal, to evaluate patient morbidity and for demonstration of good oral hygiene. Patients will be re-evaluated at 3 & 6 months post-operatively.

Test group All surgical procedure will be performed same as described in the control group except for the use of piezoelectric device for osseous resection used in this group instead of using conventional rotary instruments with carbide & diamond burs.

All patients will be prescribed an antibiotic, an anti-inflammatory/analgesic and an antiseptic mouthwash starting from the day of surgery.

PRIMARY OUTCOME

* Postoperative patient perceived outcomes
* Gain in crown length
* Change in alveolar bone level SECONDARY OUTCOME
* Stability of supracrestal gingival tissues
* Surgical time required Clinical parameters- Alginate impression will be made to provide study casts for full arch fabrication of customized probing stents.The stent will cover most of the tooth structure but away from gingival margins. The apical edge will be considered as fixed reference line for probe measurements. The following parameters will be recorded clinically and radiographically at baseline, 3 & 6months follow up period.
* Gingival index(GI), according to Löe and Silness
* Plaque index(PI), according to Silness and Löe
* Pocket probing depth(PPD)
* Free gingival margin(FGM; measured before surgery and after suturing i.e distance from stent to free gingival margin)
* Relative attachment level(RAL; measured before and after surgery i.e distance from stent to base of pocket)
* Bone level via transsulcular probing(BL-TSP; from stent under local anaesthesia before surgery and after 6months )
* Supracrestal gingival tissues will be measured by SGT=BL-TSP - FGM
* Direct bone level(DBL; before and after osseous resection measured from stent to osseous crest)
* Flap will be sutured at the level of SGT acquired post operatively.
* Postoperative pain using visual analog scale at treated site (VAS; a scale from 0-10; 0 means no pain/discomfort, 10 means maximum pain/discomfort). at these time point: 1st day, 4th day and 7th day postoperative.

All patients will be asked to fill the given format which include visual analog scale diagram ranging from 0-10 point scale.

Radiographic- Intra oral periapical radiographic evaluation of alveolar bone level will be done at baseline, after surgery and 6 months post-operatively. By taking CEJ (cement enamel junction) as a fixed reference point to alveolar bone crest, bone level will be measured at various time periods using image j software. Standardised intraoral periapical radiographs will be taken by using customized bite block with paralleling angle technique using Rinn XCP holder.

Data Collection And Methods All the data will be collected from calibrated and standardized manual periodontal probe (CP-15 UNC SE,Hu Friedy, Chicago IL). Measurements will be made at six sites on treated tooth(TT; mid-facial,mid-lingual/palatal,mesio-buccal,mesio-lingual/palatal,disto-buccal,disto-lingual/palatal)at four sites on adjacent tooth(AT; mesio-buccal, disto-buccal, mesio-lingual & disto-palatal/lingual)and at eight sites on non adjacent tooth(NA;tooth which is far from treated tooth;mesio-buccal,mesiobuccal furcation, distobuccal furcation, disto-buccal, mesio-lingual/palatal, mesio-lingual/palatal furcation, disto-lingual/palatal furcation, disto-lingual/palatal).

DATA MANAGEMENT AND STATISTICAL ANALYSIS Data recorded will be processed by standard statistical analysis. The normality of distribution of data will be examined by Shapiro Wilk test. Statistical analysis will be performed according to distribution of data. If it is in normal distribution, intra group comparison will be done by repeated ANOVA between different time points followed by paired T test between two time points and inter group comparison will be done by using Independent T test between two groups. If it is in non normal distribution, intra group comparison will be done by Wilcoxon signed rank test and inter group comparison will be done by Mann-Whitney U test. The Chi square test will be applied to analyze categoric data. Correlation and association between predictors and dependent variables will be analyzed by correlation analysis and regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60years
* plaque index(PI) <129
* gingival index(GI)<132
* short clinical abutment tooth
* crown and root fractured tooth
* tooth needed for restorative rehabilitation

Exclusion Criteria:

* Patients with systemic diseases (eg. Diabetes mellitus, hypertension, cancer patients etc.)
* Smokers
* Teeth requiring crown lengthening having adjacent tooth/teeth missing.
* Pregnant and lactating women. .Tooth mobility and furcation involvement.
* Active orthodontic therapy
* Presence of attachment loss/non restorable tooth

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative patient perceived outcomes | 7 days
  Postoperative pain using visual analog scale at treated site (VAS; a scale from 0-10; 0 means no pain/discomfort, 10 means maximum pain/discomfort)at 1st day, 4th day and 7th day postoperative..
Gain in crown length | 6 months
  Free gingival margin(FGM; measured before surgery and after suturing i.e distance from stent to free gingival margin)
Change in alveolar bone level | 6 months
  Intra oral periapical radiographic evaluation of alveolar bone level will be done at baseline, after surgery and 6 months post-operatively. By taking CEJ (cement enamel junction) as a fixed reference point to alveolar bone crest, bone level will be measured at various time periods using image j software. Standardised intraoral periapical radiographs will be taken by using customized bite block with paralleling angle technique using Rinn XCP holder.

SECONDARY OUTCOMES:
Stability of supracrestal gingival tissues | 6 months
  Supracrestal gingival tissues will be measured by SGT=BL-TSP - FGM

CONTACTS AND LOCATIONS:
Overall Officials: Shikha Tewari, MDS, Study Chair — PGIDS,ROHTAK
Locations (1):
- Shikha Tewari, Rohtak, Haryana, India